CLINICAL TRIAL: NCT05233020
Title: Robotic Assisted vs. Laparoscopic Hybrid IPOM Ventral Hernia Repair: a Prospective Randomized Study Comparing Postoperative Outcomes
Brief Title: Robotic Versus Hybrid Assisted Ventral Hernia Repair
Acronym: ROHYB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Kakela Pirjo, clinical teacher, MD, PhD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5200662
Record Dates: First submitted 2022-01-05; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Pain; Quality of Life; Recurrence
Keywords: Ventral hernia; Laparoscopy; Robot-assisted; pain
MeSH Terms: conditions — Pain; Recurrence; Hernia, Ventral

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic (Experimental): Fifteen patients undergo rVHR operation.
  Interventions: Device: robotic
- hybrid (Experimental): Fifteen patients undergo hybrid operation.
  Interventions: Device: hybrid

INTERVENTIONS:
Device: robotic — fifteen patients undergo robotic operation
  Arms: Robotic
Device: hybrid — fifteen patients undergo hybrid operation
  Arms: hybrid

SUMMARY:
Laparoscopic ventral hernia repair (LVHR) may be associated with chronic pain, seroma formation, bulging and failure to restore abdominal wall function. These outcomes are risk factors for hernia recurrence and poor quality of life (QoL). Our study evaluates whether robotic-assisted ventral hernia repair (rVHR) diminish these complications compared to LVHR with primary closure of the defect (hybrid).

DETAILED DESCRIPTION:
Thirty patients undergoing incisional ventral hernia operation with fascial defect size from 3 to 6 cm will be recruited. Fifteen patients undergo rVHR and fifteen undergo hybrid operation.The main outcome measure is postoperative pain, evaluated with visual analogue scale (VAS: 0-10) preoperatively, at 1-week, at 1-month and at 1-year. Hernia recurrence will be evaluated with ultrasound examination at 1-year and QoL using the generic SF-36 short form questionnaire preoperatively, at 1-month and at 1-year.

ELIGIBILITY:
Inclusion Criteria:

* ventral hernia size 3-6 cm

Exclusion Criteria:

* previous ventral hernia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Robotic-assisted ventral hernia repair vs hybrid. Change in pain | 1-year
  VAS scale from 0 to 10. Zero in VAS is no pain and number ten is the highest possible pain

SECONDARY OUTCOMES:
Robotic-assisted ventral hernia repair vs hybrid. Change in the social functioning status. | 1-year
  SF-36. Scale from 0 to 100. For all scales, higher scores (100) represent better function or outcome

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Käkelä, PhD, Study Director — gi -surgeon, clinical teacher; Pirjo Käkelä, PhD, Principal Investigator — gi-surgeon, clinical teacher
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No